CLINICAL TRIAL: NCT02946099
Title: Comparison of Postoperative Pain After Root Canal Instrumentation Using Reciproc and ProTaper Next in Asymptomatic Necrotic Molars: A Randomized Clinical Trial
Brief Title: Comparison Between Reciproc and Protaper Next
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ayman Abo El Enin Ahmed, Resident at Endodontic department Faculty of Oral and Dental Medecine, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: reciproc_protapernext
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Dental Pulp Necrosis
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reciproc file (Experimental): Reciproc files in reciprocating motion
  Interventions: Procedure: Reciproc files in reciprocating motion
- ProTaper Next file (Active Comparator): ProTaper Next files in continuous rotary motion
  Interventions: Procedure: ProTaper Next files in continuous rotary motion

INTERVENTIONS:
Procedure: Reciproc files in reciprocating motion — An endodontic file that works through a reciprocating motion
  Arms: Reciproc file
Procedure: ProTaper Next files in continuous rotary motion — An endodontic file that works through a continuous rotary motion
  Arms: ProTaper Next file

SUMMARY:
Comparing the postoperative pain resulting after mechanical instrumentation using Reciproc reciprocating files versus that resulting after using ProTaper Next rotary files in asymptomatic necrotic molars.

DETAILED DESCRIPTION:
Asymptomatic Necrotic molars are selected according to the eligibility and exclusion criteria and patients are then randomized to receive treatment either using Reciproc Files or ProTaper Next files. Postoperative pain is then assessed using the Numerical Rating scale 6, 12, 24 and 48 hours post-instrumentation. The tooth is then temporized and after 1 week obturation is then and post obturation pain is assessed using the Numerical Rating scale after 12 and 24 hours following obturation. The time required to complete instrumentation is also measured and compared using the two files.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular molar teeth with no pain, no response of pulp tissue to pulp testing and teeth with apical periodontitis

Exclusion Criteria:

* Patients on medication for chronic pain
* Patients with pre-operative pain.
* Patients having significant systemic disorders.
* Patients with two or more adjacent teeth requiring root canal therapy
* teeth that have vital pulp tissues, greater than grade I mobility, pocket depth greater than 5 mm, no possible restorability or previous endodontic treatment.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10-14 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Post operative pain assessed with the Numerical Rating Pain Scale | Up to 48 hours post-instrumentation
  1 to 10 Numerical Rating Pain Scale up to 48 hours post-instrumentation
Post-obturation pain assessed with the Numerical Rating Pain Scale | up to 24 hours following obturation
  1 to 10 Numerical Rating Pain Scale up to 24 hours following obturation

SECONDARY OUTCOMES:
Time required to complete instrumentation | From the completion of the access cavity preparation till the end of cleaning and shaping procedure up to 2 hours
  time required to complete instrumentation

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nekoofar MH, Sheykhrezae MS, Meraji N, Jamee A, Shirvani A, Jamee J, Dummer PM. Comparison of the effect of root canal preparation by using WaveOne and ProTaper on postoperative pain: a randomized clinical trial. J Endod. 2015 May;41(5):575-8. doi: 10.1016/j.joen.2014.12.026. Epub 2015 Feb 24. PMID 25720984
- [Background] Burklein S, Schafer E. Apically extruded debris with reciprocating single-file and full-sequence rotary instrumentation systems. J Endod. 2012 Jun;38(6):850-2. doi: 10.1016/j.joen.2012.02.017. Epub 2012 Apr 6. PMID 22595125